CLINICAL TRIAL: NCT03705559
Title: Interactions of Marijuana and Opioids: Pharmacodynamic Effects
Brief Title: Opioid and Cannabinoid Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanna Babalonis, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Shanna Babalonis, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 45017; R01DA045700 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-15 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Marijuana Usage; Opioid Use
Keywords: marijuana; opioid; opiate; cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol; Analgesics, Opioid; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double-blind, double-dummy, placebo-controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vaporized Marijuana (Experimental): Participants will receive non-therapeutic, experimental doses of active vaporized marijuana. Active marijuana will be administered once per session and will be administered via a vaporizer.
  Interventions: Drug: Vaporized Marijuana; Drug: Placebo
- Opioid Agonist (Experimental): Participants will receive non-therapeutic, experimental doses of an active opioid agonist. Active opioid agonist will be administered once per session and will be administered intranasally (snorting).
  Interventions: Drug: Opioid Agonist; Drug: Placebo
- Opioid Agonist/Marijuana Combination (Experimental): Participants will receive non-therapeutic, experimental doses of active opioid in combination with non-therapeutic, experimental doses of active vaporized marijuana. Opioid and marijuana doses will be administered once during each session. It is possible to receive both active drugs on the same day. Opioid doses will be administered intranasally; marijuana doses will be administered via vaporizer.
  Interventions: Drug: Vaporized Marijuana; Drug: Opioid Agonist
- Placebo (Placebo Comparator): Participants will receive non-therapeutic, experimental doses of placebo. Opioid doses will be administered intranasally; marijuana doses will be administered via vaporizer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaporized Marijuana — Active Marijuana administered through vaporizer
  Other Names: Cannabis; THC
  Arms: Opioid Agonist/Marijuana Combination; Vaporized Marijuana
Drug: Opioid Agonist — Active Opioid Agonist administered intranasally
  Other Names: Oxycodone
  Arms: Opioid Agonist; Opioid Agonist/Marijuana Combination
Drug: Placebo — Experimental, non-therapeutic administration of inactive opioid or marijuana dose(s)
  Arms: Opioid Agonist; Placebo; Vaporized Marijuana

SUMMARY:
This study will examine the effects of doses of marijuana/placebo and doses of opioid/placebo, alone and in combination. The primary outcomes are related to pharmacodynamic measures (subjective ratings of drug liking and other abuse-related effects; physiological outcomes) to determine the interaction effects of these compounds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 18-50
* Current non-medical use of opioids and marijuana

Exclusion Criteria:

* Physical dependence on opioids, alcohol benzodiazepines/sedative/hypnotics
* Seeking treatment for drug use
* Significant medical problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Babalonis, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Unique, randomized dose orders were created for each participant. The study utilized a within-subject design.
Groups:
- Opioid and Cannabinoid Interactions: Within subject study. Participants will receive experimental/non-therapeutic doses of active/inactive marijuana in combination experimental/non-therapeutic dose of inactive/active opioids.
Period: Overall Study
Arm/Group | Opioid and Cannabinoid Interactions
Started | 10
Placebo/Placebo | 10
THC 10mg/Placebo Opioid | 9
THC 30mg/Placebo Opioid | 10
Oxycodone 15mg/Placebo Marijuana | 9
Oxycodone 30mg/Placebo Marijuana | 9
TCH 10mg/Oxycodone 15mg | 9
TCH 10mg/Oxycodone 30mg | 9
TCH 30mg/Oxycodone 15mg | 9
TCH 30mg/Oxycodone 30mg | 9
Completed | 9
Not Completed | 1
Not completed — COVID Shut down | 1

BASELINE CHARACTERISTICS:
Population: Per protocol population. Defined as participants completing the experimental drug conditions.
Arm/Group | Opioid and Cannabinoid Interactions
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.78 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Subject-Rated Outcome - VAS Drug Liking
Description: Participants rated their subjective drug liking on a standardized VAS scale (0 to 100). Low scores mean little to no drug liking. Higher scores mean greater drug liking. Raw data transformed to peak scores.
Time Frame: This outcome (visual analog scores, scale of 0-100) was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session) and a peak score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo/Placebo: Participants will receive non-therapeutic, experimental doses of placebo. Opioid doses will be administered intranasally; marijuana doses will be administered via vaporizer.
  Placebo: Experimental, non-therapeutic administration of inactive opioid or marijuana dose(s)
- THC 10mg/Placebo Opioid; THC 30mg/Placebo Opioid: Participants will receive non-therapeutic, experimental doses of active vaporized marijuana. Active marijuana will be administered once per session and will be administered via a vaporizer.
  Vaporized Marijuana: Active Marijuana administered through vaporizer
  Placebo: Experimental, non-therapeutic administration of inactive opioid or marijuana dose(s)
- Oxycodone 15mg/Placebo Marijuana; Oxycodone 30mg/Placebo Marijuana: Participants will receive non-therapeutic, experimental doses of an active opioid agonist. Active opioid agonist will be administered once per session and will be administered intranasally (snorting).
  Opioid Agonist: Active Opioid Agonist administered intranasally
  Placebo: Experimental, non-therapeutic administration of inactive opioid or marijuana dose(s)
- TCH 10mg/Oxycodone 15mg; TCH 10mg/Oxycodone 30mg; TCH 30mg/Oxycodone 15mg; TCH 30mg/Oxycodone 30mg: Participants will receive non-therapeutic, experimental doses of active opioid in combination with non-therapeutic, experimental doses of active vaporized marijuana. Opioid and marijuana doses will be administered once during each session. It is possible to receive both active drugs on the same day. Opioid doses will be administered intranasally; marijuana doses will be administered via vaporizer.
  Vaporized Marijuana: Active Marijuana administered through vaporizer
  Opioid Agonist: Active Opioid Agonist administered intranasally
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
score on a scale | 3 (1.83) | 53.33 (10.03) | 58.89 (9.09) | 38.78 (8.29) | 35.22 (8.54) | 48.67 (10.68) | 48.00 (8.82) | 65.22 (8.02) | 72.11 (8.04)

2. Secondary Outcome: Change in Oxygen Saturation
Description: Oxygen saturation (measured as a percentage) monitored throughout each session. Raw data transformed to trough scores.
Time Frame: Oxygen saturation was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session) and a score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: percentage of oxygen saturation
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
percentage of oxygen saturation | 96.56 (0.29) | 96.44 (0.18) | 96.44 (0.18) | 96.44 (0.24) | 96.11 (0.11) | 96.22 (0.15) | 96.28 (0.30) | 95.83 (0.31) | 96.00 (0.19)

3. Secondary Outcome: Change in Respiration Rate
Description: Respiration rate (number of breaths per minute). Raw data transformed to trough scores.
Time Frame: Respiration rate was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session) and a score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: number of breaths per minute
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
number of breaths per minute | 11.89 (0.68) | 11.44 (0.56) | 12.44 (0.85) | 11.22 (0.60) | 10.22 (0.36) | 10.89 (0.35) | 10.44 (0.44) | 10.56 (0.53) | 10.89 (0.42)

4. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure (mm Hg). Raw data transformed to peak scores.
Time Frame: Blood pressure was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 8 hours per session) and a peak score was calculated across all these time intervals.
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
mm Hg | 133.56 (2.18) | 134.06 (3.50) | 140.56 (3.72) | 136.33 (3.98) | 134.33 (3.36) | 138.11 (2.87) | 139.39 (3.27) | 147.04 (5.26) | 147.56 (4.46)

5. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure (mm Hg). Raw data transformed to peak scores.
Time Frame: as for outcome 4
Population: Per Protocol population, defined as participants completing the experimental drug conditions.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
mm Hg | 89.44 (2.07) | 97.18 (2.13) | 94.92 (2.47) | 94.08 (1.59) | 91.78 (1.78) | 91.83 (2.46) | 92.67 (2.51) | 95.94 (2.22) | 98.72 (3.48)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Placebo/Placebo | THC 10mg/Placebo Opioid | THC 30mg/Placebo Opioid | Oxycodone 15mg/Placebo Marijuana | Oxycodone 30mg/Placebo Marijuana | TCH 10mg/Oxycodone 15mg | TCH 10mg/Oxycodone 30mg | TCH 30mg/Oxycodone 15mg | TCH 30mg/Oxycodone 30mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 0/9 | 1/9 | 2/9 | 2/9 | 0/9 | 3/9 | 2/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Placebo (N=9) | THC 10mg/Placebo Opioid (N=9) | THC 30mg/Placebo Opioid (N=9) | Oxycodone 15mg/Placebo Marijuana (N=9) | Oxycodone 30mg/Placebo Marijuana (N=9) | TCH 10mg/Oxycodone 15mg (N=9) | TCH 10mg/Oxycodone 30mg (N=9) | TCH 30mg/Oxycodone 15mg (N=9) | TCH 30mg/Oxycodone 30mg (N=9)
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dental Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Dryness (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Nose (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body Aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03705559/Prot_SAP_ICF_001.pdf